CLINICAL TRIAL: NCT03915158
Title: Biochemical Evaluations of Nutritional Status of Patients Before and After Bariatric and Metabolic Surgery
Brief Title: Nutritional Status of Patients Before and After Bariatric Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CMUH107-REC1-144
Record Dates: First submitted 2019-03-27; First posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Nutritional Status
MeSH Terms: interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood < 20 mL
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: bariatric surgery — sleeve gastrectomy

SUMMARY:
This study aimed at evaluating the nutritional status of vitB1, B2, B12, folate, A, D, E, Ca, Fe, Zn, Cu, and Se prior- and post- (6-Mo) the sleeve gastrectomy operation.

DETAILED DESCRIPTION:
Bariatric surgery (BS) is the most effective treatment for severe obesity and comorbidities. Among varieties of BS techniques, sleeve gastrectomy (SG) has gained in popularity worldwide. SG is a procedure involved mainly restriction combined slightly with malabsorption (deficiency in intrinsic factors for vitamin B12 absorption). Considering most patients usually have more than one micronutrients deficiency prior the surgery, the aggravated nutritional status is one of post-surgical concerns. For nutrition management, individualized biochemical assessment for micronutrients is highly recommended in guideline, but is seldom been implanted. Instead, a routine supplementation for vitamins/minerals for postoperative patients is practiced in Taiwan. This study aimed at evaluating the nutritional status of vitB1, B2, B12, folate, A, D, E, Ca, Fe, Zn, Cu, and Se prior- and post- (6-Mo) the SG operation. Subjects (n=70-100) will be recruited from patients of Body Science & Metabolic Disorders, International BMI Medical Center of CMUH. The inclusion criteria are Han Chinese, 18-65 years old, and BMI>30 who have arranged for SG operation. Written informed consent will be obtained from participants. Anthropometric data, blood samples, food (including supplements) records and medical history will be collected during the study period. We foresee this study may, not only achieve a personalized dietary plan, but also contribute to indigenous data regarding micronutrient status of obese patients.

ELIGIBILITY:
Inclusion Criteria:

* Han Chinese and Taiwanese
* BMI more than or equal to 27.5
* Surgery type is sleeve gastrectomy

Exclusion Criteria:

* Kidney dysfunction
* Mental illness
* Severe eating disorders
* Alcohol or drug abuse
* Stomach ulcers
* Redo bariatric surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from patients of Body Science & Metabolic Disorders International Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-10-31 (Estimated); Study Completion 2019-10-31 (Estimated)

PRIMARY OUTCOMES:
Change of Nutritional status | pre-surgery and 6 months after surgery
  Blood sample will be collected and used to determine nutritional status which will measured by laboratory biochemical test.

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Min Chao, PhD, Principal Investigator — Department of Nutrition, China Medical University
Locations (1):
- China Medical University, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lin CH, Liao WL, Wu CC, Shaw HM, Hsu WL, Lu YC, Yang JS, Huang CK, Chao PM. Nutritional Status of Obese Taiwanese Before Bariatric-Metabolic Surgery and Their Serum 25-Hydroxyvitamin D Concentrations for Maximal Suppression of Parathyroid Hormone. Obes Surg. 2020 Oct;30(10):3940-3946. doi: 10.1007/s11695-020-04759-y. Epub 2020 Jul 8. PMID 32638247